CLINICAL TRIAL: NCT07136831
Title: "Short-term Outcome of Patients From Rural Versus Urban Communities Undergoing Primary Percutaneous Coronary Intervention for ST-Elevation Myocardial Infarction"
Brief Title: "Short-term Outcome in STEMI Patients Undergoing Primary PCI: A Comparative Study Between Rural and Urban Communities at Assiut University."
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Ali Khallaf, Principal Investigator, Assiut University
Other Study IDs: STEMI-PPCI-RURALURBAN-ASU25
Record Dates: First submitted 2025-07-28; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: MACE; In STEMI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months

INTERVENTIONS:
Device: Primary Percutaneous Coronary Intervention (PPCI) — A catheter-based invasive procedure used to open blocked coronary arteries in patients presenting with ST-elevation myocardial infarction (STEMI).

SUMMARY:
this study aims to assess the short-term (3-month) clinical and echocardiographic outcomes of primary PCI among STEMI patients from rural versus urban areas in Upper Egypt. A special focus will be placed on identifying predictors of MACE. The findings may offer valuable insight into optimizing STEMI care pathways and support the development of regional STEMI networks across Egypt.

DETAILED DESCRIPTION:
ST-segment elevation myocardial infarction (STEMI) is a life-threatening condition that requires urgent reperfusion therapy, with primary percutaneous coronary intervention (PCI) being the gold standard of care. While PCI significantly reduces complications and improves survival, access to this intervention remains unequal, particularly between rural and urban populations

According to the latest census definitions, a rural area is characterized by:A population of fewer than 5,000,A population density of less than 400 persons per square kilometer,And more than 25% of the male working population engaged in agriculture.

Rural patients often experience delayed diagnosis, limited access to PCI-capable centers, and prolonged ischemic times. These factors contribute to poorer clinical outcomes, including higher rates of reinfarction, heart failure, and mortality. In contrast, urban residents typically have faster access to specialized cardiac care and more efficient treatment pathways.

In Upper Egypt, this urban-rural gap is particularly pronounced, with rural patients facing substantial logistical and systemic challenges in receiving timely PCI. Although efforts have been made to expand PCI access nationwide, there remains a lack of localized data comparing short-term outcomes-particularly major adverse cardiovascular events (MACE)-between rural and urban STEMI patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adults aged ≥18 years. 2. Confirmed diagnosis of ST-segment elevation myocardial infarction (STEMI) based on ECG and cardiac biomarkers.

  3. Underwent primary percutaneous coronary intervention (PCI) within the study period.

  4. Known and verified residential address classified as rural or urban based on official definitions (e.g., UK or WHO classification).

  5. Informed consent obtained

Exclusion Criteria:

1. Non-STEMI or unstable angina cases.
2. Patients who received fibrinolytic therapy instead of PCI.
3. Transfer from another facility after more than 12 hours of symptom onset.
4. Patients with previous revascularization (e.g., CABG or PCI within the last 6 months).
5. Incomplete clinical data or unknown residential location.

   -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients Confirmed diagnosis of ST-segment elevation myocardial infarction (STEMI) based on ECG and cardiac biomarkers.
Sampling Method: Probability Sample
Enrollment: 162 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of major adverse cardiovascular events (MACE) among STEMI patients undergoing primary percutaneous coronary intervention (PCI), | 3 month
  Unite of measurement : Number of patients experiencing MACE (% of total)

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/36044196
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6425633/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9677036/